CLINICAL TRIAL: NCT06390020
Title: Mindfulness-Based Stress Reduction for People High on the Personality Trait Sensory Processing Sensitivity: A Mixed Methods Study
Brief Title: Mindfulness-Based Stress Reduction (MBSR) for People High on the Personality Trait Sensory Processing Sensitivity: A Mixed Methods Study
Acronym: MindSens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL84880.091.23
Record Dates: First submitted 2024-03-20; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-03

CONDITIONS: Sensory Processing Sensitivity
Keywords: Sensory processing sensitivity; Highly sensitive person; Mindfulness-based stress reduction; Mindfulness; Depression; Anxiety; Stress; Self-regulation
MeSH Terms: conditions — Depression; Anxiety Disorders; Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants instructed not to partake in any (similar) mindfulness or meditation training.
- MBSR training (Experimental)
  Interventions: Other: MBSR

INTERVENTIONS:
Other: MBSR — The MBSR training spans eight weeks and follows a standardized protocol. It consists of eight weekly sessions, each lasting 2.5 hours, a single 6-hour silent day, and daily home exercises. Additionally, the program incorporates personalized psychoeducation on high sensory processing sensitivity, covering its characteristics, scientific foundations, its relation with stress-related symptoms, and why mindfulness might be helpful.
  Arms: MBSR training

SUMMARY:
This study investigates the efficacy of MBSR training in alleviating stress-related symptoms among individuals with high sensory processing sensitivity. Participants will be randomly allocated to either the MBSR group or the control group.

The primary hypothesis is that participants in the MBSR group, relative to control group, will have lower depression-anxiety-stress scores post-intervention, after controlling for baseline scores. The secondary hypothesis is that in the MBSR group, relative to control group, other mental health, physical health and well-being outcomes, as well as potential mindfulness mechanisms will also improve, after controlling for baseline scores.

ELIGIBILITY:
Inclusion Criteria:

* Participant has high sensory processing sensitivity (screened for by the Highly Sensitive Person Scale (HSPS) with a mean score of ≥4.4)
* Participant is 18 years or older
* Participant is proficient in Dutch
* Participant lives near the location where the MBSR training takes place (up to about 30km from Nijmegen)
* Participant is able to travel to location of the MBSR training for all sessions
* Participant is available on the scheduled times of the MBSR sessions (or not available for one session with exception of the silent day)

Exclusion Criteria:

* Participant has a severe psychological condition (e.g. psychotic or suicidal)
* Participant has followed mindfulness or meditation training (~eight-week program) within the previous five years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Post-intervention in self-reported depression, anxiety, and stress | Baseline, Post-intervention at approximately 3 months
  Measured by the Depression, Anxiety and Stress Scale (DASS-21). It has 21 items assessed on a four-point Likert scale (0-3) with a total score ranging from 0 to 63. There are three subscales (Depression, Anxiety and Stress), with each seven items and subscale scores ranging from 0 to 21. The main outcome will be the total score, which is doubled to match the scores of the full version (DASS-42). A higher score indicates more severe symptoms of depression, anxiety, and/or stress.

SECONDARY OUTCOMES:
Change from Baseline to Post-intervention in self-reported well-being | Baseline, Post-intervention at approximately 3 months
  Measured by the Mental Health Continuum - Short Form (MHC-SF). It has 14 items assessed on a six-point Likert scale (0-5) with a total score ranging from 0 to 70. There are three subscales: Emotional well-being (3 items), Social well-being (5 items), and Psychological well-being (6 items). Score combinations across these subscales can be used to distinguish between the following subgroups: flourishing, moderate, and languishing. Higher scores indicate a better well-being.
Change from Baseline to Post-intervention in self-reported burnout symptoms | Baseline, Post-intervention at approximately 3 months
  Measured by the Burnout Assessment Tool - Short Form (BAT-12). It has 12 items assessed on a five-point Likert scale (1-5) with a mean total score ranging from 1 to 5. There are four subscales: Exhaustion, Mental Distance, Emotional Impairment, and Cognitive Impairment (3 items each). Mean subscale scores range from 1 to 5. Higher scores indicate more severe burnout symptoms.
Change from Baseline to Post-intervention in self-reported physical symptoms | Baseline, Post-intervention at approximately 3 months
  Measured by the Cohen - Hoberman Inventory of Physical Symptoms (CHIPS). It has 33 items assessed on a five-point Likert scale (0-4) with a total score of 0 to 132. A higher score indicates more severe physical symptoms.
Change from Baseline to Post-intervention in self-reported overstimulation | Baseline, Post-intervention at approximately 3 months
  Measured by the Multi-Modal Evaluation of Sensory Sensitivity (MESSY). It has 30 items assessed on a five-point Likert scale (1-5) with a total score of 30 to 150. There are seven subscales Multisensory Sensitivity (7 items), Visual Sensitivity (5 items), Auditory Sensitivity (5 items), Tactile Sensitivity (3 items), Chemosensory Sensitivity (4 items), Sensitivity to environmental temperature (3 items), and Motion Sensitivity (3 items). Mean subscale scores range from 1 and 5. Higher scores indicate more overstimulation symptoms.
  The three secondary outcomes listed above, in addition to this one, can be categorized into outcomes pertaining to mental and physical health as well as well-being.
Change from Baseline to Post-intervention in self-reported mindfulness | Baseline, Post-intervention at approximately 3 months
  Measured by the Five Facet Mindfulness Questionnaire - Short Form (FFMQ-SF). It has 24 items assessed on a five-point Likert scale (1-5) with a total score ranging from 24 to 120. There are five subscales: Observing (4 items), Describing (5 items), Acting with awareness (5 items), Non-judging (5 items), and Nonreactivity (5 items) with subscale scores ranging from 4 to 20 for Observing and from 5 to 25 for the others. Higher scores indicate more mindfulness.
Change from Baseline to Post-intervention in self-reported attention regulation | Baseline, Post-intervention at approximately 3 months
  Measured by the Attention Control Scale (ACS). It has 20 items assessed on a four-point Likert scale (1-4) with a total score ranging from 20 to 80. There are two subscales: Attention Focusing (9 items) with a subscale score ranging from 9 to 36 and Attention Shifting (11 items) with a subscale score ranging from 11 to 44. Higher scores indicate more attention regulation.
Change from Baseline to Post-intervention in self-reported strategies for cognitive emotion regulation | Baseline, Post-intervention at approximately 3 months
  Measured by the Cognitive Emotion Regulation Questionnaire - Short Form (CERQ-SF). It has 18 items assessed on a five-point Likert scale (1-5). This study uses eight of in total nine subscales (and 16 items) with two items each: four adaptive strategy subscales: (Putting into perspective, Positive reappraisal, Positive refocusing, and Refocus on planning), and four less adaptive strategies (Self-blame, Other-blame, Rumination, and Catastrophizing). Subscale scores range from 2 to 10 and higher scores indicate more of that emotion regulation strategy.
Change from Baseline to Post-intervention in self-reported body awareness | Baseline, Post-intervention at approximately 3 months
  Measured by the Multidimensional Assessment of Interoceptive Awareness - 2 (MAIA-2). It has 37 items assessed on a six-point Likert scale (0-5). There are eight subscales: Noticing (4 items), Not Distracting (6 items), Not-Worrying (5 items), Attention Regulation (7 items), Emotional Awareness (5 items), Self-Regulation (4 items), Body Listening (3 items), and Trusting (3 items) with mean subscale scores ranging from 0 to 5. Higher scores indicate more of that body awareness aspect.
Change from Baseline to Post-intervention in self-reported self-compassion | Baseline, Post-intervention at approximately 3 months
  Measured by the Self-Compassion Scale - Short-Form (SCS-SF). It has 12 items assessed on seven-point Likert scale (1-7) with a total score ranging from 12 to 84. There are six subscales: Self-Kindness, Self-Judgement, Common Humanity, Isolation, Mindfulness, and Over-Identified with two items each. Subscale scores range from 2 and 14. Higher scores indicate more self-compassion.
  The four secondary outcomes listed above, in addition to this one, can be categorized into outcomes pertaining to potential mindfulness mechanisms.
Change from Baseline to Post-intervention in self-reported sensory processing sensitivity | Baseline, Post-intervention at approximately 3 months
  Measured by the Sensory Processing Sensitivity Questionnaire - Short Form (SPSQ-SF). It has 26 items assessed on a seven-point Likert scale (1-7) with a total score ranging from 26 to 182. There are six subscales: Sensory sensitivity to subtle internal and external stimuli (4 items), Social affective sensitivity (5 items), Aesthetic sensitivity (3 items), Sensory comfort (5 items), Sensory discomfort (4 items), and Emotional and physiological reactivity (5 items). The first four subscales make up the positive dimension and the last two subscales the negative dimension. Subscale scores and dimension scores are derived by adding up the relevant items. Higher scores indicate more sensory processing sensitivity aspects.
Perceived facilitators, barriers, effects, and mechanisms of participating in the MBSR training | Post-intervention at approximately 3 months
  Semi-structured interview, participant observer

CONTACTS AND LOCATIONS:
Overall Officials: Anne Speckens, prof. dr., Principal Investigator — Radboudumc, Centre for Mindfulness; Corina Greven, prof. dr., Principal Investigator — Donders Centre for Cognitive Neuroimaging
Locations (1):
- The Radboudumc Center for Mindfulness, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Greven CU, Lionetti F, Booth C, Aron EN, Fox E, Schendan HE, Pluess M, Bruining H, Acevedo B, Bijttebier P, Homberg J. Sensory Processing Sensitivity in the context of Environmental Sensitivity: A critical review and development of research agenda. Neurosci Biobehav Rev. 2019 Mar;98:287-305. doi: 10.1016/j.neubiorev.2019.01.009. Epub 2019 Jan 9. PMID 30639671